CLINICAL TRIAL: NCT05555563
Title: Effect of MTAD on The Outcome of Primary Root Canal Treatment: A Randomized Controlled Trial
Brief Title: Effect of MTAD on The Outcome of Primary Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Berkcan Yıldız, Research Assistant, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDH-2019-12197
Record Dates: First submitted 2022-06-27; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Dental Pulp Disease; Periapical Diseases; Tooth, Nonvital
Keywords: Apical periodontitis; Biopure MTAD; Randomized Clinical Trial
MeSH Terms: conditions — Dental Pulp Diseases; Periapical Diseases; Tooth, Nonvital; Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Root canal instrumentation was performed using the Reciproc Blue (VDW, Munich) #50/0.5 file. During instrumentation of the root canals, irrigation was applied with 10 mL 2.5% NaOCl using side-vented needles. The final irrigation in Control group was applied with 5 ml of 17% EDTA solution and 5 ml of distilled water. The root canals were dried with sterile paper points and were filled with cold lateral condensation technique using AH Plus root canal sealer and gutta percha. Then the cavity entry was restored with composite (Solarex, GC Corparation, Tokyo, Japan) and radiography was taken. The pre-treatment and 24-month follow-up radiographs of teeth, were prepared as a Power Point presentation and the change in periapical radiolucency was assessed according to PAI scores Teeth with a PAI≤ 2 score and clinically asymptomatic were considered 'healthy' in the radiographic evaluation, while teeth with a PAI≥ 3 and/or clinically symptomatic were considered 'failure'.
- MTAD irrigation (Experimental): Root canal instrumentation was performed using the Reciproc Blue (VDW, Munich) #50/0.5 file. During instrumentation of the root canals, irrigation was applied with 10 mL 2.5% NaOCl using side-vented needles. The final irrigation in MTAD group was applied 5 ml MTAD (n=50) and 5 ml of distilled water. The root canals were dried with sterile paper points and were filled with cold lateral condensation technique using AH Plus root canal sealer and gutta percha. Then the cavity entry was restored with composite (Solarex, GC Corparation, Tokyo, Japan) and radiography was taken. The pre-treatment and 24-month follow-up radiographs of teeth, were prepared as a Power Point presentation and the change in periapical radiolucency was assessed according to PAI scores Teeth with a PAI≤ 2 score and clinically asymptomatic were considered 'healthy' in the radiographic evaluation, while teeth with a PAI≥ 3 and/or clinically symptomatic were considered 'failure'.
  Interventions: Other: MTAD irrigation

INTERVENTIONS:
Other: MTAD irrigation — Final irrigation protocol was performed using 5 ml MTAD (n=50).
  Other Names: Aysin Dumani
  Arms: MTAD irrigation

SUMMARY:
The aim of this clinical study was to compare the radiographic outcome of a root canal treatment with or without use of MTAD after 24 months recall. This in vivo study was a prospective, single-center; single blinded, parallel, and randomized clinical trial. The study protocol was approved by the Ethics Committee of Cukurova University Faculty of Medicine.

One hundred patients with a noncontributory medical history presented to the Department of Endodontics of the University of Cukurova Faculty of Dentistry between October 2019 and February 2020 were selected according to inclusion and exclusion criteria. All selected teeth were single-rooted, maxillary and mandibular incisors, canines or premolars that were asymptomatic (no preoperative pain, swelling or acute endodontic or periodontal abscess). All pulps were nonvital and did not respond to cold testing. All patients were aged between 18 and 65 years, had no systemic diseases or allergies tolocal anaesthetic agents, had not previously received any endodontic treatment and had no radiographic evidence of periapical bone loss. Pregnant and breast-feeding women and patients taking analgesic, anti-inflammatory or antibiotic medications during the 7 days prior to the beginning of treatment were also excluded. All patients were informed that they were to be included in a clinical trial and their consent was obtained.The initial periapical radiographs of the patients were taken with the digital imaging system Digora Optime (Soredex, Tuusula, Finland) by long-cone paralleling technique with a film holder (Endo Rh plus; Indusbello, Londrina, PR, Brazil), the vitality of the pulp was evaluated by an electronic vitalometer (Analytic Technology Corp., Redmond, WA, USA) and confirmed by the absence of bleeding from the endodontic access cavity.

For both maxillary and mandibular teeth, local infil-tration anaesthesia was achieved using 2 mL articaine hydrochloride with 1:200 000 adrenaline (Maxicaine; VEM Ilac, Istanbul, Turkey). Endodontic access preparations were performed using diamond round burs. After the canals were visible, patency was checked with a K-file (VDW GmbH, Munich, Germany), and a dental dam was placed to isolate the tooth. The working length (WL) was determined with an electronic apex locator (Raypex 6,VDW) and accepted when all 3 green bars were reached. In addition, the canal length was confirmed by a periapical radiograph, and the apex locator was accepted as correct in situations where the two did not match. Root canal instrumentation was performed using the Reciproc Blue (VDW, Munich) #50/0.5 file. During instrumentation of the root canals, irrigation was applied with 10 mL 2.5% NaOCl using side-vented needles (NaviTips, 30 gauge; Ultradent, South Jordan, UT, USA). The final irrigation in Control group was applied with 5 ml of 17% EDTA solution and 5 ml of distilled water. In the MTAD group, final irrigation was done with 5 mL of MTAD and 5 mL of distilled water. Side-vented needles were placed 1 mm shorter than the working length, and 5 ml of solution was given in 2 minutes. The root canals were dried with sterile paper points and were filled with cold lateral condensation technique using AH Plus root canal sealer (Dentsply Maillefer, Cologne, Germany) and gutta percha (President Dental, Duisburg, Germany). Then the cavity entry was restored with composite (Solarex, GC Corparation, Tokyo, Japan) and radiography was taken. Patients were invited to follow-up sessions at 6, 12, 18, and 24 months and were radiographically and clinically assessed. Many patients missed their follow-up appointments due to the covid 19 pandemic. The follow-up radiographs performed by long-cone paralleling technique with a film holder. The pre-treatment and 24-month follow-up radiographs of teeth, were prepared as a Power Point presentation (Microsoft ® Corporation, Redmond, WA) and the change in periapical radiolucency was assessed according to PAI scores of five categories; 1. Normal apical periodontium 2. Small changes in bone structures 3. Change in bone structure with mineral loss 4. Periodontitis with well-defined radiolucent area 5. Severe periodontitis with exacerbating features. Teeth with a PAI≤ 2 score and clinically asymptomatic were considered 'healthy' in the radiographic evaluation, while teeth with a PAI≥ 3 and/or clinically symptomatic were considered 'failure'.

DETAILED DESCRIPTION:
This randomized controlled clinical trial was conducted to evaluate radiographic periapical repair after endodontic treatment using 5 mL of MTAD and 5 mL of distilled water (MTAD group) or 5 ml of 17% EDTA solution and 5 ml of distilled water (Control group) irrigation in single-rooted teeth with apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* No systemic diseases
* No history of taking analgesics in the previous seven days or other drugs prior to presenting for treatment
* All selected teeth were necrotic, single root teeth with a periapical lesion ( 2>PAI ≤5 mm)

Exclusion Criteria:

* Systemic and/or periodontal disease
* Allergy to local anesthetic agents and/or histrory of intolerance to nonsteroidal anti-inflammatory drugs;
* Requirement for antibiotic prophylaxis
* Open tooth apex
* Pacemaker use
* Women were pregnant or breastfeeding status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Healing of periapical lesions by radiographic findings according to periapical index (PAI). | Long-term follow-up evaluation in 24 months. Each patient will recall for an appointment and the periapical status of the tooth will be evaluated by periapical radiograph.
  The periapical index (PAI) is structured scoring system for categorization of radiographic features of apical lesion. It is based on a visual scale of periapical periodontitis severity and was built upon a classical study of histological-radiological correlations. It is a five-point ordinal scale as listed below: 1. Normal apical periodontium. 2. Small changes in bone structures. 3. Change in bone structure with mineral loss. 4. Periodontitis with well-defined radiolucent area. 5. Severe periodontitis with exacerbating features.and MTAD group

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Torabinejad M, Cho Y, Khademi AA, Bakland LK, Shabahang S. The effect of various concentrations of sodium hypochlorite on the ability of MTAD to remove the smear layer. J Endod. 2003 Apr;29(4):233-9. doi: 10.1097/00004770-200304000-00001. PMID 12701769
- [Result] Mozayeni MA, Javaheri GH, Poorroosta P, Ashari MA, Javaheri HH. Effect of 17% EDTA and MTAD on intracanal smear layer removal: a scanning electron microscopic study. Aust Endod J. 2009 Apr;35(1):13-7. doi: 10.1111/j.1747-4477.2007.00111.x. PMID 19452675
- [Result] Verma N, Sangwan P, Tewari S, Duhan J. Effect of Different Concentrations of Sodium Hypochlorite on Outcome of Primary Root Canal Treatment: A Randomized Controlled Trial. J Endod. 2019 Apr;45(4):357-363. doi: 10.1016/j.joen.2019.01.003. Epub 2019 Mar 1. PMID 30827769
- [Result] Huumonen S, Orstavik D. Radiographic follow-up of periapical status after endodontic treatment of teeth with and without apical periodontitis. Clin Oral Investig. 2013 Dec;17(9):2099-104. doi: 10.1007/s00784-013-0926-2. Epub 2013 Feb 5. PMID 23385425
- [Result] Ng YL, Mann V, Rahbaran S, Lewsey J, Gulabivala K. Outcome of primary root canal treatment: systematic review of the literature - part 1. Effects of study characteristics on probability of success. Int Endod J. 2007 Dec;40(12):921-39. doi: 10.1111/j.1365-2591.2007.01322.x. Epub 2007 Oct 10. PMID 17931389
- [Result] Orstavik D, Kerekes K, Eriksen HM. The periapical index: a scoring system for radiographic assessment of apical periodontitis. Endod Dent Traumatol. 1986 Feb;2(1):20-34. doi: 10.1111/j.1600-9657.1986.tb00119.x. No abstract available. PMID 3457698
- [Result] Tosun S, Karataslioglu E, Tulgar MM, Derindag G. Fractal analysis and periapical index evaluation of multivisit nonsurgical endodontic retreatment: A retrospective study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2022 Feb;133(2):245-251. doi: 10.1016/j.oooo.2021.08.016. Epub 2021 Aug 30. PMID 34556458

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT05555563/Prot_SAP_ICF_000.pdf